CLINICAL TRIAL: NCT00856037
Title: A Phase I Study of Weekly Doxorubicin and Oral Topotecan for Patients With Relapsed or Refractory Small Cell Lung Cancer (SCLC)
Brief Title: Topotecan Hydrochloride and Doxorubicin Hydrochloride in Treating Relapsed or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0508-08-FB; NCI-2009-01308 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (doxorubicin hydrochloride, topotecan hydrochloride) (Experimental): Patients receive doxorubicin hydrochloride IV over 3-5 minutes on day 6 of course 1 and on days 6, 13, and 20 of courses 2-5. Patients also receive topotecan hydrochloride PO on days 1-5. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Topotecan Hydrochloride — Given PO
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)

SUMMARY:
This phase I trial studies the side effects and best dose of topotecan hydrochloride when given together with doxorubicin hydrochloride in treating patients with small cell lung cancer (SCLC) that has come back after a period of improvement (relapsed) or has not responded to treatment (refractory). Drugs used in chemotherapy, such as topotecan hydrochloride and doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Doxorubicin hydrochloride may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving topotecan hydrochloride and doxorubicin hydrochloride may be a better treatment for small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and efficacy, in terms of clinical disease benefit, (complete or partial response and stable disease with stable or improved quality of life scores) of combination of oral topotecan (topotecan hydrochloride) when given with weekly doxorubicin (doxorubicin hydrochloride) in patients with SCLC.

II. Determine the dose limiting toxicity of oral topotecan when given with weekly doxorubicin in patients with SCLC.

SECONDARY OBJECTIVES:

I. Estimate topoisomerase I and II levels in peripheral blood mononuclear cells and correlate with presence or absence of grades 3 and 4 hematological toxicity.

II. Estimate topoisomerase I and II levels in peripheral blood mononuclear cells and correlate with efficacy.

OUTLINE: This is a dose-escalation study of topotecan hydrochloride.

Patients receive doxorubicin hydrochloride intravenously (IV) over 3-5 minutes on day 6 of course 1 and on days 6, 13, and 20 of courses 2-5. Patients also receive topotecan hydrochloride orally (PO) on days 1-5. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of small cell lung cancer (SCLC)
* Have received at least one prior chemotherapy regimen for SCLC
* Primarily refractory or relapsed disease
* Measurable or evaluable disease: measurable disease in 2 dimensions on imaging studies performed within 4 weeks of starting treatment
* Greater than 2 weeks since last treatment (chemotherapy or radiation) provided subject has recovered from side effects of treatment prior to the study
* Karnofsky score >= 70; (Eastern Cooperative Oncology Group [ECOG] 0-2)
* No active secondary malignancy; patients with other prior malignancies will be included, provided they have been disease-free for at least five years
* Patients with adequately treated basal cell or squamous cell carcinoma of the skin, adequately treated non-invasive carcinomas will be eligible
* White blood cell (WBC) count >= 3,500/mm^3 within 7 days prior to starting treatment, OR
* Absolute neutrophil count (ANC) >= 1,500/ul within 7 days prior to starting treatment
* Platelet count >= 100,000/mm^3 within 7 days prior to starting treatment
* Serum creatinine less than 1.5 times the upper limits of normal within 7 days prior to starting treatment
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 1.5 times the upper limits of normal within 7 days prior to starting treatment in the absence of liver metastasis; in the presence of liver metastasis serum AST and ALT less than or equal to 5.0 times the upper limits of normal within 7 days prior to starting treatment
* Serum alkaline phosphatase less than 2.5 times the upper limits of normal within 7 days prior to starting treatment in the absence of liver metastasis; in the presence of liver metastasis serum alkaline phosphatase less than or equal to 5.0 times the upper limits of normal within 7 days prior to starting treatment
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study; (no childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)
* Non-pregnant and non-nursing; men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on the study
* Able to return for treatment and follow-up as specified in the protocol
* Able to give informed consent

Exclusion Criteria:

* Known hypersensitivity to any component of topotecan or doxorubicin or other required drugs in the study
* Any co morbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Ejection fraction below the lower limit of normal (< 50%)
* Uncontrolled intercurrent illnesses including, but not limited to unstable angina or uncontrolled cardiac arrhythmia, chronic liver disease, complete left bundle branch block, obligate use of a cardiac pacemaker, ST depression of > 1 mm in two or more leads and/or T wave inversions in two or more contiguous leads, congenital long QT syndrome, history of or presence of significant ventricular or atrial tachyarrhythmias, clinically significant resting bradycardia (< 50 beats per minute), corrected QT (QTc) > 480 ms on screening electrocardiogram that could jeopardize the patient?s ability to receive the chemotherapy described in the protocol safely
* Women who are pregnant (confirmed by a serum pregnancy test in females of reproductive potential) or breast-feeding; women of child-bearing potential and sexually active males must be advised to take precautions to prevent pregnancy during treatment (unless the subject or subject?s partner(s) is sterile (i.e. women who have had a hysterectomy or have been post-menopausal for at least twelve consecutive months) or remain abstinent, men and women of reproductive potential must agree to use TWO of the following forms of birth control every time they have sex throughout the study and for up to 3 months following discontinuation of study drug: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicidal, intrauterine device (IUD), or surgical sterilization while participating in this study; hormonal birth control methods are not permitted
* Inability to co-operate with the requirements of the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02-02 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the next lowest dose level below where greater than or equal to 2/3 or 3/6 patients experience dose limiting toxicities in cohorts of 5 different doses by National Cancer Institute Common Toxicity Criteria version 3.0 | Up to 6 weeks (after 2 courses)
  The actual rates of dose limiting toxicities per dose cohort will be presented when applicable.

SECONDARY OUTCOMES:
Changes in topoisomerase I and II levels in peripheral blood mononuclear cells | Baseline to up to week 16
  The changes over time will be described and correlated with hematological toxicity and efficacy. Mean change and standard deviation over time will be computed and when possible change in topoisomerase levels over time will be compared between patients developing grade 4 hematological toxicities versus others (no toxicity or grades 1-3) or between patients developing grades 3-4 non-hematological toxicities versus others (no toxicity or grades 1-2) or between patients who responded (complete response, partial response, stable disease) versus no response or progressed using non-parametric tests.
Overall response rate | Up to 15 weeks (after 5 courses)
  complete or partial response and stable disease
Changes in quality of life levels | Up to 16 weeks
  Measured by standard instruments and compared when possible between patients who responded versus nonresponders.

CONTACTS AND LOCATIONS:
Overall Officials: Apar Ganti, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States